CLINICAL TRIAL: NCT00529828
Title: Health Effects of CLA Versus Industrial Trans Fatty Acids in Healthy Volunteers (CLARINeT-Study)
Brief Title: Health Effects of CLA Versus Industrial Trans Fatty Acids
Acronym: CLARINeT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: VU University of Amsterdam (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NL15599.081.07
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Healthy
Keywords: CLA; Industrial trans fatty acids; Oleic acid; Controlled dietary trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Consumption of CLA enriched food

SUMMARY:
The knowledge of the health effects of CLA on the human body is limited. However, CLA supplements are sold over the counter in several countries and various techniques are used to increase the content of CLA in food.

The CLARINeT study will be performed to investigate the effect of CLA on blood lipoproteins, inflammatory markers, blood pressure and insulin status in human volunteers relative to industrial trans fatty acids and to oleic acid.

DETAILED DESCRIPTION:
It will be a double-blind randomized multiple cross-over trial with 3 treatments:

* CLA;
* Industrial trans fatty acids (as a positive control);
* Oleic acid (Cis 18:1, the monounsaturated fatty acid in unhydrogenated vegetable oils) as a reference fat.

Each volunteer receives each diet for three weeks, in random order, for a total of 9 weeks. Three weeks is sufficient to reach new stable lipoprotein levels.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* healthy

Exclusion Criteria:

* serum total cholesterol >= 6,5 mmol/L
* serum triglycerides > 2,3 mmol/L
* chronic diseases (such as diabetes, cardiovascular disease, kidney and liver dysfunction)
* use of cholesterol lowering medication
* use of blood pressure lowering medication
* high alcohol intake
* BMI > 30
* pregnant and lactation women
* unusual dietary requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Total cholesterol
HDL cholesterol
LDL cholesterol
Apo B
Triglycerides

SECONDARY OUTCOMES:
Insulin status markers : HOMA; QUICKY
Inflammatory markers: C-RP; IL-6; E-selectin; MCP-1; s-TNF-R1; s-TNF-R2; IFg
Fatty acid composition of cholesteryl esters and erythrocytes
proteomics
iso-prostanes
blood pressure and heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Brouwer, Dr., Principal Investigator — VU University of Amsterdam; Martijn Katan, Prof. Dr., Principal Investigator — VU University of Amsterdam
Locations (1):
- Wageningen University, Division of Human Nutrition, Wageningen, Netherlands

REFERENCES:
- [Derived] Smit LA, Katan MB, Wanders AJ, Basu S, Brouwer IA. A high intake of trans fatty acids has little effect on markers of inflammation and oxidative stress in humans. J Nutr. 2011 Sep;141(9):1673-8. doi: 10.3945/jn.110.134668. Epub 2011 Jul 13. PMID 21753062
- [Derived] Wanders AJ, Brouwer IA, Siebelink E, Katan MB. Effect of a high intake of conjugated linoleic acid on lipoprotein levels in healthy human subjects. PLoS One. 2010 Feb 3;5(2):e9000. doi: 10.1371/journal.pone.0009000. PMID 20140250